CLINICAL TRIAL: NCT00880282
Title: A Phase I Study of IMC-A12 (Anti-Insulin-Like Growth Factor-I Receptor Monoclonal Antibody) in Combination With CCI-779 (Temsirolimus) in Pediatric Patients With Recurrent or Refractory Solid Tumors
Brief Title: Cixutumumab and Temsirolimus in Treating Younger Patients With Solid Tumors That Have Recurred or Not Responded to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01910; NCI-2011-01910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0813; CDR0000639150; ADVL0813 (Other: Children's Oncology Group); ADVL0813 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — cixutumumab; temsirolimus; Sirolimus

ARMS (1):
- Treatment (cixutumumab, temsirolimus) (Experimental): Patients receive cixutumumab IV over 60 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 25 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Drug: temsirolimus; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cixutumumab — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of cixutumumab when given together with temsirolimus in treating younger patients with solid tumors that have recurred or not responded to treatment. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and recommended Phase II dose of IMC-A12 (anti-insulin growth factor-1 receptor monoclonal antibody) (cixutumumab) administered as an intravenous infusion once weekly in combination with CCI-779 (temsirolimus) administered intravenously once weekly to children with refractory solid tumors.

II. To define and describe the toxicities of IMC-A12 in combination with temsirolimus administered on this schedule.

III. To characterize the pharmacokinetics of IMC-A12 in combination with temsirolimus in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of the combination of IMC-A12 and temsirolimus within the confines of a Phase I study.

II. To assess the biologic activity of IMC-A12 by assessing: changes in insulin-like growth factor receptor (IGFR) expression and phosphorylation and insulin-receptor expression and phosphorylation in peripheral blood mononuclear cells (PBMNC).

III. To assess the biological activity of temsirolimus by measuring levels of phosphorylated (phosphor)-ribosomal protein S6 kinase, 70kDa, polypeptide 1 (S6K1), phosphor-protein kinase B (AKT), phosphor-eukaryotic translation initiation factor 4 gamma, 1 (eIF4G) in PBMNC.

IV. To assess the incidence of IGFR expression as well as mechanistic target of rapamycin (mTOR) pathway activation in recurrent or refractory solid tumors of childhood.

OUTLINE:

Patients receive cixutumumab intravenously (IV) over 60 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 25 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of serum or cerebrospinal fluid (CSF) alpha-fetoprotein or beta-human chorionic gonadotropin (HCG); slides or tissue blocks from either initial diagnosis or relapse must be available for central review
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; note: neurologic deficits in patients with central nervous system (CNS) tumors must have been clinically stable for a minimum of 1 week prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: must not have received within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
  * Hematopoietic growth factors: at least 7 days since the completion of therapy with a growth factor that supports platelet or white cell number or function
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent; at least 6 weeks must have elapsed since prior therapy that includes a monoclonal antibody; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Radiation therapy (XRT): >= 2 wks for local palliative XRT (small port); >= 3 months must have elapsed if prior total-body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; >= 6 wks must have elapsed if other substantial bone marrow (BM) radiation
  * Stem cell transplant or rescue: no evidence of active graft vs. host disease and >= 2 months must have elapsed since transplant
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * 0.6 mg/dL (for patients 1 year of age)
  * 0.8 mg/dL (for patients 2 to 5 years of age)
  * 1 mg/dL (for patients 6 to 9 years of age)
  * 1.2 mg/dL (for patients 10 to 12 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (for patients 13 to 15 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (for patients >= 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum albumin >= 2 g/dL
* Patients with seizure disorder may be enrolled if receiving non-enzyme inducing anticonvulsants and well controlled
* Prothrombin time (PT) and international normalized ratio (INR) < 1.2 x ULN
* Random or fasting blood glucose within the upper normal limits for age; if the initial blood glucose is a random sample that is outside of the normal limits, then a follow-up fasting blood glucose can be obtained and must be within the upper normal limits for age
* Serum cholesterol and serum triglyceride levels must be < grade 2
* All patients and/or their parents or legal guardians must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of the study and for 3 months after the last dose of IMC-A12.
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anticancer agents are not eligible
* Patients receiving insulin or growth hormone therapy are not eligible
* Patients must not be receiving enzyme-inducing anticonvulsants
* Patients must not be receiving any of the following potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers or inhibitors: erythromycin, clarithromycin, ketoconazole, azithromycin, itraconazole, grapefruit juice or St. John's wort
* Patients receiving warfarin for the purpose of systemic anticoagulation are not eligible; use of low-dose warfarin for maintaining patency of central venous catheters is allowed
* Patients who have an uncontrolled infection are not eligible
* Patients with known type I or type II diabetes mellitus are not eligible
* Patients with known bone marrow involvement are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients who have received prior monoclonal antibody therapy targeting IGF-1R or temsirolimus are not eligible
* Patients with history of allergic reactions attributed to compounds of similar chemical; or biologic composition to IMC-A12 or temsirolimus are not eligible
* Patients must not have had major surgery for 6 weeks prior to enrollment on the study; patients with history of recent minor surgical procedures (vascular catheter placement, bone marrow evaluation, laparoscopic surgery) will be eligible

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose and recommended phase II dose based on the incidence of dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days
Toxicities as assessed by the NCI CTCAE version 4.0 | Up to 30 days after the last dose of treatment
Pharmacokinetics (PK) of cixutumumab | At end of infusion, at 1, 3, 6, and 24 hours, days 1, 4, 8, 15, 22, and 28 (of course 1), and days 15 and 28 (of course 2)
  The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Pharmacokinetics of temsirolimus | At end of infusion, at 15 and 30 minutes, at 1, 3, 6, and 24 hours, days 1, 4, 7, and 28 (of course 1), and days 15 and 28 (course 2)
  The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

SECONDARY OUTCOMES:
Disease response according to Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 4 years
  Reported descriptively.
Change IGFR and insulin receptor expression | From baseline to up to 28 days (of course 1)
  Summary statistics and descriptive plots will be generated for IGFR expression. The changes will be assessed using paired t-test or Wilcoxon matched pairs signed rank sum test when appropriate.
Change in levels of S6K1, AKT, eIF4G, and associated phosphoproteins | From baseline to up to 28 days (of course 1)
  Summary statistics and descriptive plots will be generated. The changes will be assessed using paired t-test or Wilcoxon matched pairs signed rank sum test when appropriate.
Incidence of IGFR expression as well as mTOR pathway activation | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — Children's Oncology Group
Locations (23):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Childrens Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mark O Hatfield-Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec